CLINICAL TRIAL: NCT00934479
Title: The Intestinal Microecology in Chronic Constipation
Brief Title: Intestinal Microecology in Chronic Constipation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, John K. DiBaise, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-001281
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Other Constipation; Irritable Bowel Syndrome
Keywords: Chronic Constipation; Constipation Predominant Irritable Bowel Syndrome; Intestinal Microecology
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Subjects (No Intervention): Healthy subjects completed a baseline 1-week diary of stool and defecatory characteristics, fasting breath for hydrogen and methane and a stool sample for pyrosequencing. Otherwise, the healthy subjects received no intervention.
- Constipated Subjects (Experimental): Subjects with constipation included those with chronic constipation (CC) and those with constipation predominant irritable bowel syndrome (C-IBS). They completed a baseline 1-week diary of stool and defecatory characteristics, fasting breath for hydrogen and methane and a stool sample for pyrosequencing.
  Following baseline test and because of differences in the FDA-approved dosing for the 2 subtypes of chronic constipation, the CC subjects received open-label lubiprostone 24 mcg orally twice daily for 4 weeks; while the C-IBS subjects received open-label lubiprostone 8 mcg orally twice daily for 4 weeks.
  Following the 4-weeks treatment with lubiprostone, they completed another stool diary, fasting breath test, and stool sample for pyrosequencing.
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — Following the initial stool and breath collections and because of differences in the FDA-approved dosing for the 2 subtypes of chronic constipation, (that is, chronic constipation (CC) versus constipation due to irritable bowel syndrome (C-IBS), the CC subjects received open-label lubiprostone 24 mcg orally twice daily for 4 weeks; while the C-IBS subjects received open-label lubiprostone 8 mcg orally twice daily for 4 weeks.
  Other Names: Amitiza
  Arms: Constipated Subjects

SUMMARY:
The purpose of this study is to determine whether the bacteria normally present in the bowels are different in people with constipation and to see what effect the treatment with the Food and Drug Administration (FDA) - approved drug, lubiprostone, has on these bacteria.

DETAILED DESCRIPTION:
Chronic constipation is a common condition with a heterogeneous pathophysiology and resulting clinical manifestations. Recent evidence in the literature and collected in our laboratory confirm that there are differences in the gut microbiota between healthy individuals and those with a variety of disorders (e.g., inflammatory bowel disease, irritable bowel syndrome and obesity) suggesting that the development of certain disorders may be determined by the composition of the gut microbiota. Existing evidence warrants further investigation of the role of the microbial ecology of the human gut in constipation and an exploration of modification of the gut microbiota as a means to treat constipation by its actions on the colonic metabolism of nutrient substrates to alter colonic transit and fluid fluxes.

The proposed research will exploit our proven capability to use high-throughput molecular genomic techniques to define the intestinal microbiome in order to help define the role of the gut microbiota in chronic constipation and will explore the potential value of altering the microbiota as a management strategy in constipation. The linkage of high-throughput genomic analyses with cause-and-effect understanding of how the gut microbiota affects bowel function may lead to a reliable means to manage the gut microbiota with the intent to prevent and/or treat constipation. The immediate goals of this project are to expand on existing information about the microbial ecology in the human intestines focusing on its relationship with constipation using molecular microbiological techniques and to assess the effects on the gut microorganisms resulting from the use of the FDA-approved medication, lubiprostone. Lubiprostone is a member of a novel therapeutic class called prostones and is an orally active, bicyclic fatty acid that selectively acts on type 2 chloride channels to stimulate chloride secretion which induces a net increase in luminal fluid secretion. Unlike antibiotic, probiotic and prebiotic agents, it has no known direct effects on the gut microbiota. It is FDA-approved for the treatment of chronic constipation in men and women and for women with constipation-predominant IBS (C-IBS). The rationale for using lubiprostone to modify the gut microbiota stems from the use of similar strategies for controlling recalcitrant small intestinal bacterial overgrowth (i.e., altering fluid fluxes in the gut lumen).

We believe that this research will greatly improve our understanding of the role that the gut microbiota play in the development of constipation and potentially lead to new strategies with which to combat this common problem.

ELIGIBILITY:
Inclusion Criteria for Healthy Subjects:

1. Fewer than 3 bowel movements/day and more than 3 bowel movements/week without the need for significant straining with defecation or frequent sensation of incomplete evacuation after defecation
2. Absence of current or chronic gastrointestinal symptoms

Inclusion Criteria for Chronic Constipation Subjects:

1. Meet Rome III criteria for chronic functional constipation
2. Colonoscopy within the previous 10 years for subjects ≥ 50 years of age

Inclusion Criteria for Constipation-Predominant IBS Patients:

1. Meet Rome III criteria for C-IBS
2. Colonoscopy within the previous 10 years for subjects ≥ 50 years of age

Exclusion Criteria:

1. Prior gastrointestinal surgery that altered the anatomy of the esophagus, stomach, or small/large intestine (exceptions include appendectomy and cholecystectomy)
2. Gastrointestinal, cardiovascular, endocrine, renal, or other chronic disease likely to affect gastrointestinal motility (e.g., uncontrolled diabetes mellitus)
3. Females of childbearing age who are not practicing birth control and/or are pregnant or lactating (a urine pregnancy test will be performed on female subjects prior to lubiprostone use)
4. Significant untreated psychiatric disease
5. History of hypersensitivity reaction or intolerance to lubiprostone
6. Inability to stop antibiotics, probiotics, and fiber supplements 1 month prior to stool sample collection
7. Inability to stop proton pump inhibitors, histamine 2 receptor antagonists, prokinetic agents, narcotic analgesic agents, laxatives, and anticholinergic agents 2 weeks prior to stool sample collection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Identification of specific microorganisms associated with chronic constipation in comparison to healthy subjects and those with C-IBS | 5 weeks

SECONDARY OUTCOMES:
Evaluate changes in the gut microbiota after lubiprostone treatment in the chronic constipation subjects and those with C-IBS | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John K. DiBaise, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Kang DW, DiBaise JK, Ilhan ZE, Crowell MD, Rideout JR, Caporaso JG, Rittmann BE, Krajmalnik-Brown R. Gut microbial and short-chain fatty acid profiles in adults with chronic constipation before and after treatment with lubiprostone. Anaerobe. 2015 Jun;33:33-41. doi: 10.1016/j.anaerobe.2015.01.005. Epub 2015 Jan 21. PMID 25617726